CLINICAL TRIAL: NCT07120854
Title: Evaluation of a Decision Analysis Model in a Decision Aid for Fracture Prevention in Postmenopausal Women: Randomized Clinical Trial.
Brief Title: Evaluation of a Decision Analysis Model in the DASH-Osteo Decision Aid.
Acronym: DASH-Osteo
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Institut Catala de Salut (Other Government); Servicio Madrileño de Salud, Madrid, Spain (Other); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24/202-P
Record Dates: First submitted 2025-07-28; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporotic Fractures; Diphosphonates; Fracture Risk Assessment
Keywords: postmenopausal; osteoporotic fractures; primary prevention
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporotic Fractures | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Decision aid plus decision analysis model (Experimental): Participants in this group will use DASH-Osteo decision aid plus the information in plain language, provided by a decision analysis model which will include the utilities provided by the same participants in the web- based tool, and will make a shared decision with their healthcare professional.
  Interventions: Other: Decision aid with decision analysis model
- Decision aid only (Experimental): Participants in this group will use DASH-osteo decision and will make a shared decision with their healthcare professional.
  Interventions: Other: Decision aid alone
- Control (Active Comparator): Participants in this group will make a decision according to centre's usual practice
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Decision aid with decision analysis model — Women will use the web version of the decision aid tool. They will have a supporting video to help them how to navigate the tool during. They will be able to access the tool through a specific link that will be shared with them by their central research team via e-mail. Each woman is expected to use the web tool and select her preferences (utilities) regarding different health conditions (e.g. hip fracture). The results of the exercises will be received automatically at the central level (by institutional e-mail to the researcher responsible for the data a PDF file will be sent from the web). The research team at the central level will apply the decision analysis model, using information on the baseline fracture risk and preferences of each participant entered into the tool. The results of the decision analysis model will be delivered to the women directly by e-mail in plain language, so that they can make the final decision together with their general practitioner in a second visit.
  Arms: Decision aid plus decision analysis model
Other: Decision aid alone — Participants will use the web tool. They will have a supporting video to help them how to navigate the tool during. They will be able to access the tool through a specific link that will be shared with them by the central research team via e-mail. Each woman is expected to navigate through the different functions of the web tool, at home or at a time other than the medical visit, and select her preferences (utilities) with respect to different health conditions (e.g. hip fracture). The women in this group would decide whether or not to take the pharmacological treatment based on the information provided by the tool but without the results of the decision analysis model described for the intervention group. Subsequently, those who wished to do so would make a final decision together with their physician at a second visit.
  Arms: Decision aid only
Other: Usual Care — Women in this group will receive standard clinical practice, without the use of the shared decision support tool or the decision analysis model or any other support. At the end of the visit, their physician will provide them with a link to access the assessment questionnaires.
  Other Names: Usual practice
  Arms: Control

SUMMARY:
Fragility fractures, often caused by low bone mineral density, are a major health concern for postmenopausal women. One way to prevent these fractures is by taking medication, but deciding whether to start treatment can be difficult due to potential risks and side effects.

This study will test a web-based tool designed to help women make informed decisions about fracture prevention treatment. The tool provides information about the benefits and risks of treatment. Some women in the study will also receive additional support through a decision analysis report, which helps weigh different factors when making a choice.

The study will examine whether using this tool improves decision-making, increases confidence in making a choice, and enhances satisfaction with the decision. It will also explore what factors influence women's decisions and at what level of risk they choose to start treatment.

By understanding how decision aids impact choices, researchers aim to improve the way healthcare providers support patients in making informed decisions about their health.

DETAILED DESCRIPTION:
Open-label, randomized, open-label, multicenter, three parallel arms, controlled clinical trial. It will be carried out in primary care centers belonging to the Autonomous Communities of Madrid and Catalonia.

The participants will be recruited in the medical consultation, by their family doctor, who will assess the fulfillment of the inclusion criteria a priori and according to eligibility, will offer the woman to participate in the study, informing her about the nature of the research. The informed consent form will be signed online, and the inclusion criteria will be verified by the participant herself when accessing the tool. Participation will be voluntary and does not entail economic incentives for the participants.

Random assignment will be simple following a 1:1:1 ratio to each group. To avoid possible contamination bias, randomization will be performed at the physician level, so that each professional will be randomized to one of the intervention groups so that he/she will apply exclusively one of the study's interventions to all the participants he/she recruits. Due to the characteristics of the interventions it will not be possible to blind the interveners and participants. After randomization, only the data analysts will be blinded to the randomization sequence. The central research team will primarily contact participants via email to send the decision aid tool link and questionnaire links. They will also follow up to ensure the completion of all data provided by the participants.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women older than 50 years
* No medical history of fragility fractures
* With or without a BMD measurement performed
* Having been considered candidates to pharmacological treatment prevention for fragility fractures.
* A 10 year fracture risk assessment according to FRAX for Major fracture >5%.

Exclusion Criteria:

* women with a history of fragility fracture
* being treated with bisphosphonates or other osteoporosis drugs (except for vitamin D and calcium supplements
* suffer from serious concomitant pathologies (cancer, chronic renal insufficiency, etc.)
* women under permanent treatment with glucocorticoids.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — As fragility fracture risk is higher in older women due to their estrogen decrease. We will include only postmenopausal women.
Enrollment: 114 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | Decisional conflict will be measured one time up to 26 weeks, after participant use of the web-based tool.
  We will use the Decisional conflict scale (O'Connor 1998, updated 2010), to evaluate the uncertainty and the decision-making conflict across participants. It is a 16-item scale. IItems are summed, then multiplied by 25.
  Scoring goes from 0 (low decisional conflict) to 100 (high decisional conflict). Patients with a total score >38 tend to delay decisions, whereas those with ≤ 25 tend to make decisions(1, 2)
  1. O'Connor AM. Validation of a Decisional Conflict Scale. Med Decis Making [Internet]. 1995 Feb;15(1):25-30. Available from: http://dx.doi.org/10.1177/0272989X9501500105
  2. Bunn H, O'Connor A. Validation of Client Decision-Making Instruments in the Context of Psychiatry. Can J Nurs Res [Internet]. 1996;28(3):13-27. Available from: https://pubmed.ncbi.nlm.nih.gov/8997937/

SECONDARY OUTCOMES:
Decision self-efficacy | Decision-Self-efficacy scale will be applied, up to 26 weeks, after using the decision aid tool.
  Participants, self-confidence with the decision, will be measured with the Decision Self-efficacy scale (O'Connor 1995, updated 2002) a 11-item 5-point validated scale. Items are summed, then divided by 11 and then multiplied by 25.
  Scores range from 0 ("extremely low self-efficacy") to 100 ("extremely high"). The scale is reliable and has been validated in different populations (1, 2).
  1. Bunn H, O'Connor A. Validation of Client Decision-Making Instruments in the Context of Psychiatry. Can J Nurs Res [Internet]. 1996;28(3):13-27.
  2. Galiana L, Sánchez-Ruiz J, Gómez-Salgado J, Larkin PJ, Sansó N. Validation of the Spanish Version of the Five-Item General Self-Efficacy (GSE) Scale in a Sample of Nursing Students: Evidence of Validity, Reliability, Longitudinal Invariance and Changes in General Self-Efficacy and Resilience in a Two-Wave Cross-Lagged Panel Model. Nurse Educ Pract [Internet]. 2024 Jan;74:103865.
Participant satisfaction with the decision process | Satsfaction will be assessed up to 26 weeks, after participant's second visit with their physician.
  We will measure participants satisfaction with the decision satisfaction scale from Holmes-Rovner 1996 (SWD). SWD scale is a 6-item validated scale scoring from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater satisfaction with the decision (1, 2, 3
  1. Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, et al. Patient Satisfaction with Health Care Decisions: The Satisfaction with Decision Scale. Med Decis Making [Internet]. 1996 Feb;16(1):58-64. doi.org/10.1177/0272989X9601600114
  2. Wills CE, Holmes-Rovner M. Preliminary Validation of the Satisfaction With Decision scale with Depressed Primary Care Patients. Health Expect [Internet]. 2003 Jun;6(2):149-59. doi.org/10.1046/j.1369-6513.2003.00220.x
  3. Chabrera C, Areal J, Font A, Caro M, Bonet M, Zabalegui A. Versión española de la Satisfaction With Decision scale: adaptación transcultural, validez y fiabilidad. Enferm Clin [Internet]. 2015 May;25(3):117-23. dx.doi.org/10.1016/j.enfcli.2015.0

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No